CLINICAL TRIAL: NCT05340634
Title: Evaluation of the Efficacy of the Combination of Antioxidants Metionac for the Modulation of Metabolic and Endocrine Parameters in Patients With Polycystic Ovary Syndrome: A Prospective Randomized Study.
Brief Title: Evaluation of Metionac for the Modulation of Metabolic and Endocrine Parameters in Patients With PCOS.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Margan Biotech (Industry)
Collaborators: Grupo CINUSA (Centros de Investigación en Nutrición y Salud S.L.) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOP-DIET
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Contraceptive (Active Comparator): Drospirenone 4 mg once a day for 6 months
  Interventions: Drug: Oral contraceptive
- Oral Contraceptive + Food supplement Metionac (Experimental): Drospirenone 4 mg once a day and Metionac twice daily (200 mg S-adenosylmethionine, 100 mg N-acetylcisteine, 75 mg alpha lipoid acid and 0,65 Vitamin B6) for 6 months
  Interventions: Dietary Supplement: Metionac; Drug: Oral contraceptive
- Food supplement MetioNac (Other): Metionac twice daily (200 mg S-adenosylmethionine, 100 mg N-acetylcisteine, 75 mg alpha lipoid acid and 0,65 Vitamin B6) for 6 months
  Interventions: Dietary Supplement: Metionac

INTERVENTIONS:
Dietary Supplement: Metionac — Metionac is a food suplement composed by 200 mg of SAMe, 100 mg of NAC, 75 mg of ALA and 0,65 mg of vitamin B6 per tablet for 6 months
  Arms: Food supplement MetioNac; Oral Contraceptive + Food supplement Metionac
Drug: Oral contraceptive — Drospirenone 4 mg once a day
  Arms: Oral Contraceptive; Oral Contraceptive + Food supplement Metionac

SUMMARY:
Evaluate the efficacy of the combination of antioxidants ALA, NAC, Vit. B6 and SAMe as a dietary supplement, in the improvement of metabolic and endocrine parameters and clinical manifestations of PCOS.

DETAILED DESCRIPTION:
The investigators will explain the study to all patients who meet the inclusion and exclusion criteria during the study period. After signing the informed consent patients will be randomized 1:1 to oral contraceptive 4 mg drospirenone once daily or oral contraceptive 4 mg drospirenone + combination of 200 mg S-adenosylmethionine, 100 mg N-acetylcisteine, 75 mg Alpha lipoid acid and 0,65 mg vitamin B6 (Metionac) twice daily. Patients for whom oral contraceptive is not indicated will be enrolled in third study group of Metionac twice daily. 2 study visits will be carried out, Baseline (Visit 0) and after 6 months therapy (Visit 1).

ELIGIBILITY:
Inclusion Criteria:

1. Women newly diagnosed with PCOS with at least 2 of the following symptoms:

   * Oligo/Anovulation < 21 or > 35 days > 90 days (any cycle) < 8 periods / year
   * Hyperandrogenism (clinical symptoms or laboratory results)
   * Polycystic ovary morphology (NHMRC guideline): In any ovary:

     20 follicles* and/or ovarian volume greater than or equal to 10ml and no corpus luteum, cysts or dominant follicles

     *number of follicles per ovary measuring 2-9 mm
2. > 18 years old
3. Overweight defined as BMI>25
4. Normal prolactin levels
5. Women with altered coagulation factors or a personal history of thromboembolism for whom OAC is contraindicated (they will be included in the control group without randomization)
6. Written inform consent

Exclusion Criteria:

1. Diabetic women
2. Adrenal enzyme deficiency and/or other endocrine disease
3. Pregnant or lactating women.
4. Women under treatment with SNRIs (serotonin reuptake inhibitors)
5. Other serious illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Mean BMI at 6 Months | 6 months
  Evolution of Body Mass Index in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Insuline level at 6 Months | 6 months
  Evolution of Insuline level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Glucose level at 6 Months | 6 months
  Evolution of Glucose level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Triglycerides at 6 Months | 6 months
  Evolution of Triglycerides level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean HDL at 6 Months | 6 months
  Evolution of high-density lipoprotein (HDL) cholesterol level in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean LDL at 6 Months | 6 monhts
  Evolution of low-density lipoprotein (LDL) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean AST at 6 months | 6 months
  Evolution of aspartate aminotransferase (AST) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean ALT at 6 months | 6 months
  Evolution of alanine aminotransferase (ALT) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean GGT at 6 months | 6 months
  Evolution of gamma glutamyltransferase (GGT) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Bilirubin at 6 Months | 6 months
  Evolution of total and free bilirubin level in patients with PCOS after 6 months therapy

SECONDARY OUTCOMES:
Change from Baseline in the Mean 17 beta estradiol at 6 months Translate from: English volume_up 20 / 5,000 Translation results Change from baseline in the Mean 17 beta estradiol at 6 Months | 6 months
  Evolution of 17 beta estradiol level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean 17 hydroxy progesterone at 6 months Translate from: English volume_up 20 / 5,000 Translation results Change from baseline in the Mean 17 beta estradiol at 6 Months | 6 months
  Evolution of 17 hydroxy progesterone level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean LH at 6 months Translate from: English volume_up 20 / 5,000 Translation results Change from baseline in the Mean 17 beta estradiol at 6 Months | 6 months
  Evolution of luteinizing hormone (LH) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean FSH at 6 months Translate from: English volume_up 20 / 5,000 Translation results Change from baseline in the Mean 17 beta estradiol at 6 Months | 6 months
  Evolution of follicle-stimulating hormone (FSH) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Testosterone at 6 months | 6 months
  Evolution of testosterone level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Androstenedione at 6 months | 6 months
  Evolution of androstenedione level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean DHEA at 6 months | 6 months
  Evolution of Dehydroepiandrosterone (DHEA) level in patients with PCOS after 6 months therapy
Change from Baseline in the Mean TSH at 6 months | 6 months
  Evolution of thyroid stimulating hormone (TSH) level in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean Homocysteine at 6 months | 6 months
  Evolution of homocysteine (HC) level in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean HOMA-IR at 6 months | 6 months
  Evolution of HOMA insulin resistance level in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean Hb A1c at 6 months | 6 months
  Evolution of hemoglobin A1c in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean SHBG at 6 months | 6 months
  Evolution of sex hormone binding globulin in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean Hirsutism score at 6 months | 6 months
  Evolution of hirsutism score measured by Ferriman - Gallwey scale in patients with PCOS after 6 months therapy. The Ferriman-Gallwey scale for hirsutism. A score of 1 to 4 is given for nine areas of the body. A total score less than 8 is considered normal, a score of 8 to 15 indicates mild hirsutism, and a score greater than 15 indicates moderate or severe hirsutism. A score of 0 indicates absence of terminal hair.
Change from Baseline in the Mean Acne self-assessment score at 6 months | 6 months
  Evolution of acne self assessed from 1 to 10 (1 minimum severity, 10 maximum severity) in acne severity level in 3 areas: face, neck, back in patients with PCOS after 6 months therapy.
Change from Baseline in the Mean Alopecia score at 6 months | 6 months
  Evolution of alopecia using Ludwig scale in patients with PCOS after 6 months therapy. The Ludwig hair loss scale illustrates progressive hair loss patterns in women. It ranges from I to III. Stage I begins with thinning on the top of the head. In stage II the scalp starts to show. All of the hair at the crown of the head may be lost when the hair loss progresses to stage III.Stage I begins with thinning on the top of the head. In stage II the scalp starts to show. All of the hair at the crown of the head may be lost when the hair loss progresses to stage III.
Change from Baseline in the Proportion of patients with irregular menstrual cycle at 6 months | 6 months
  Regularization of irregular menstrual cycle in patients with PCOS after 6 months therapy
Change from Baseline in the Mean Migraine score at 6 months | 6 months
  Evolution of migraine score using Migraine Disability Assessment test (MIDAS) in patients with PCOS after 6 months. The MIDAS score is derived as the sum of missed days due to a headache over a 3-month period in the three domains: school work or work for pay; household work or chores; and family, social, and leisure activities. The four-point grading system for the MIDAS questionnaire is as follows:
  • Grade 1 (scores ranging from 0 to 5): little or no disability Grade 2 (scores ranging from 6 to 10): mild disability Grade 3 (scores ranging from 11 to 20): moderate disability Grade 4 (21 or greater): severe disability.
Change from Baseline in the Mean QoL score at 6 months | 6 months
  Evolution of quality of life score using Health-Related Quality of Life Questionnaire for women with Polycystic Ovary Syndrome (adapted from PCOSQ qustionnaire) in patients with PCOS after 6 months therapy. The PCOS HRQL questionnaire represents a new measure for women with PCOS and includes five domains: emotional, body hair, infertility, weight, and menstrual problems. A shorten version with 19 questions was used. It ranges from 0 (no impact on quality of life to 114 maximum negative impact in the patient´s quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Quironsalud San José, Madrid, Spain